CLINICAL TRIAL: NCT00131612
Title: An Investigation of the Effect of the Promoter Polymorphism in the Glucuronosyltransferase 2B7 Using Epirubicin Clearance and the Ratios of Epirubicin and Epirubicinol Glucuronide to Epirubicin
Brief Title: An Investigation of the Effect of the Promoter Polymorphism in the Glucuronosyltransferase 2B7 in Patients on Breast Cancer Treatment
Status: Terminated | Type: Observational
Why Stopped: did not apply for ethics renewal
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: BR-01-0031 / 17027
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: adjuvant therapy; epirubicin; uridine glucuronosyl/transferase 2B7; pharmacogenetics
MeSH Terms: conditions — Breast Neoplasms | interventions — FEC protocol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: FEC 100 — 5-fluoruracil, epirubicin and cyclophosphamide every three weeks for six treatments

SUMMARY:
For many years scientists and cancer researchers have been trying to find out why some people benefit more from anti-cancer medications than other people who receive the same amount and same kind of medications. Current studies suggest that inherited characteristics might explain these differences. Height and eye color are examples of characteristics that have been inherited from parents. Studies suggest that people might also inherit genetic differences in how their bodies break down medications. When a person receives an anti-cancer medication, it is broken down by the liver into smaller parts or by-products. To try to understand more about how people's bodies break down anti-cancer medications, the researchers are studying the by-products (called metabolites) of epirubicin in the blood of people who are taking this medication as part of their breast cancer treatment.

DETAILED DESCRIPTION:
Epirubicin is an anthracycline that is widely used in breast cancer, stomach and esophageal cancer. Despite epirubicin being the 4'-epi-isomer of doxorubicin, epirubicin undergoes substantially different metabolism compared to doxorubicin. The majority of epirubicin is metabolized to glucuronides, 78.0% to epirubicin glucuronide and 19.3% to epirubicinol glucuronide and only 0.2% epirubicin is metabolized to epirubicinol. Doxorubicin is primarily metabolized to aglycones or doxorubicinol but not to glucuronides. There is substantial variability in epirubicin metabolism with the mean clearance of 84.6 L/h and a standard deviation of 63.5. A study by Hu et al showed epirubicin metabolism correlated with response. In this study they showed patients with nasopharyngeal cancer treated with epirubicin were more likely to relapse if they rapidly metabolized epirubicin. A study by Robert et al raises the possibility that the differences in epirubicin metabolism are determined by genetic differences. They showed a bimodal distribution in the ratio of epirubicin glucuronides to epirubicin. As well this study showed that low glucuronidation were more likely to respond to epirubicin than patients who had a high ratio of epirubicin glucuronides to epirubicin. Innocenti et al has shown that epirubicin is metabolized to its glucuronides by uridine glucuronosyltransferase 2B7 (UGT2B7). The same study showed a strong correlation between the formation of morphine-6-glucuronide and the glucuronidation of epirubicin in human liver microsomes. The researchers have recently discovered a single nucleotide polymorphism in the enhancer region of UGT 2B7. Patients who were homozygous for this polymorphism tended to have lower ratios of morphine-6-glucuronide to morphine. The researchers suspect that this T to C polymorphism decreases the transcription of UGT 2B7 and this is the basis of the decreased glucuronidation. Given the strong correlation between the metabolism of morphine and epirubicin in human liver microsomes the researchers suspect that this polymorphism may be responsible for the variability in epirubicin metabolism. Previous work has documented an overlapping bimodal distribution in the ratio of epirubicin glucuronides but they did not examine whether genetic polymorphisms were responsible for this. This study will examine the effect of this polymorphism on the metabolism of epirubicin. If a relationship exists between this polymorphism and epirubicin metabolism this may allow more accurate dosing of this important chemotherapeutic agent.

Objectives:

To determine in patients receiving adjuvant intravenous FEC chemotherapy (5-Fluoruracil 500 mg/m2, epirubicin 100 mg/m2, Cyclophosphamide 500 mg/m2) given every 3 weeks whether the newly discovered SNP at position -161 T to C is responsible for the variability in epirubicin metabolism.

Participants:

Patients receiving adjuvant FEC chemotherapy. Patients can not have pre-existing liver disease other than Gilbert's syndrome. In patients with a history of liver disease, liver transaminases must be less than 3 times the upper limit of normal and bilirubin less than the upper limit of normal. Patients must be >/= 18 years of age.

Eligible patients will be enrolled into the study after written informed consent is obtained. Baseline characteristics including age, weight, renal function, liver function, concurrent medications and ethnic origin will be obtained from the medical chart or patient. The patient chart will be reviewed periodically for hematological and nonhematological toxicity. Outcome data such as recurrence and time of recurrence will be obtained from the chart.

Sample Size:

Medical oncologists consider a significant difference in drug clearance to be 15%. Epirubicin's clearance is 84.6 L/h with a standard deviation of 63.5. The researchers have calculated a sample size to have an 80% power to detect a 15% difference. Assuming epirubicin's average clearance is comprised of three separate groups, which is the hypothesis, the researchers would need 29 patients from each genotype to show a 15% difference between the mean clearance of different genotypes assuming a coefficient of variation of 20%. The known polymorphism at amino acid residue 268 has an allele frequency of 50%. This allele was in complete linkage disequilibrium with the new SNP at position -160 in the previous study of morphine. Therefore the researchers would need approximately 120 patients to produce 30 T/T, 60 T/C and 30 C/C.

ELIGIBILITY:
Inclusion Criteria:

* Receiving adjuvant or neoadjuvant FEC100

Exclusion Criteria:

* Elevated bilirubin
* Abnormal liver or kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross Cancer Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2002-01; Primary Completion 2005-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada